CLINICAL TRIAL: NCT07008950
Title: Self-efficacy and Knowledge (SEEK) Trial to Improve Sexual Reproductive Health and Well-being for Syrian Refugee Women and Girls in Lebanon
Acronym: SEEK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: World Health Organization (Other); Elrha (Other)
Responsible Party: Principal Investigator, Shadi Saleh, Professor and Founding Director of the Global Health Institute, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SBS-2023-0310; 78689 (Other: ELRHA)
Record Dates: First submitted 2025-02-28; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Mental Health Care; Sexual Health Quality of Life; Family Planning Services
Keywords: sexual health; reproductive health; psychosocial support; wellbeing; RCT; Lebanon; Refugees; Girls and young women

STUDY DESIGN:
Intervention Model Description: This study will report on a community based RCT in which syrian refugee women and girls aged 15-24 recruited from 2 PHCs in Lebanon were randomly allocated into control and experimental groups. The aim is to examine changes in key outcomes of sexual reproductive health, family planning, and wellbeing as a result of receiving the WHO-developed integrated intervention package. The experimental group will receive the intervention package by attending 8 sessions on this topic over a period of 8 weeks. The control group will not receive the intervention package.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group receiving SEEK intervention (Experimental): Participants randomly assigned to the experimental group will be further randomly assigned to 16 subgroups of no more than 12 participants per groups to receive the SEEK integrated intervention package on sexual reproductive health, family planning, and wellbeing.
  Interventions: Other: The Self-Efficacy and Knowledge Trial
- Control group not receiving SEEK intervention (No Intervention)

INTERVENTIONS:
Other: The Self-Efficacy and Knowledge Trial — The intervention is composed on 8 sessions given over a period of 8 weeks covering topics of emotional regulation, communication, problem management, decision making, self-efficacy and others in relation to sexual reproductive health, family planning, and wellbeing. The intervention package will be delivered by trained non-specialists with at least 12 years of formal education. The package will be administered once a week for a duration of 90 minutes.
  Arms: Group receiving SEEK intervention

SUMMARY:
This community-based randomized controlled trial (RCT) aims to evaluate a low-resource/low-intensity integrated sexual reproductive health (SRH) and wellbeing intervention package. It will be delivered in Primary Healthcare Centres (PHCs) in a rural area in Lebanon to Syrian refugee women and girls aged 15-24.

DETAILED DESCRIPTION:
Use and access to sexual and reproductive health (SRH) services are often inadequate and limited among adolescent girls and young refugee women in humanitarian settings. This is attributed to an array of factors including: limited health literacy, lack of knowledge on where and how to access services, limited availability of services, and gender norms. Further, the nature of humanitarian settings often poses additional mental health pressures because of limited safety, political instability, gender-based violence (GBV), and dire socio-economic and living conditions, among others. This is especially true for the Eastern Mediterranean Region (EMR), which hosts the largest number of humanitarian crises in the world, thus rendering the provision of SRH and psychosocial support (PSS) services in humanitarian settings highly compromised.

The proposed research aims to evaluate the impact of a WHO-developed low-intensity/low-resource psychosocial support (PSS) SRH-integrated intervention package on the use of selected SRH services, primarily family planning as well as well-being among Syrian adolescent girls and young women refugees, aged 15-24 years, in Lebanon. The research will adopt a community-based randomized controlled trial (RCT) design to evaluate the effectiveness of the PSS-SRH integrated intervention package on the use of selected SRH services as well as mental well-being. The RCT will be accompanied by a rigorous process evaluation during intervention implementation to assess intervention fidelity, attrition, dose and satisfaction, as well as to capture key lessons based on intervention implementation to inform global scale-up in different humanitarian settings.

This intervention is expected to be easily integrated into existing primary healthcare settings and specifically to improve selected SRH service use, leading to improved SRH outcomes and reduced SRH-related risks, and ultimately better wellbeing among refugee women and girls. Findings of this RCT are also expected to inform key stakeholders and better guide decision making for such interventions in humanitarian settings.

ELIGIBILITY:
Inclusion Criteria:

-

The target population of the study are Syrian adolescent girls and young women refugees (age 15-24 years) residing in Beqaa governorate in Lebanon. Participants will be included in the study if they meet the following inclusion criteria:

1. are currently married and between the ages of 15 - 24 years,
2. completed an average stay in Lebanon for a minimum of 6 months,
3. are willing to take part in the study as indicated by them signing an informed consent (for young women 18 years of age or older) or through a legal guardian consent form and written assent for adolescents' girls between 15 and 17,
4. have none of the exclusion criteria listed below upon screening.

Exclusion Criteria:

Participants will be excluded from the study if they meet any of the following criteria:

1. are currently pregnant and/or lactating,
2. have reported chronic health problems interfering with the ability to follow the intervention protocol,
3. have high levels of anxiety and/or depression as well as suicidal ideations and/or attempts upon screening and/or a current diagnosis of a severe mental illness, or undergoing mental health treatment.

   -

Ages: 15 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Only females assigned at birth who identify as women
Enrollment: 485 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Family Planning Use | From enrollement until 3 months post intervention delivery
  Improvement in family planning use among the EG compared to the CG at 3 months post intervention. This will be measured using the Pan Arab-Family Health (PAPFAM) survey. This is a descriptive tool with values indicating use or no use of family planning services. It is not scored, but rather yields un-scored percentages. Higher percentages may mean worse or better outcomes depending on the question.

SECONDARY OUTCOMES:
Anxiety and Depression Measure | From enrollment until 3 months post intervention
  Improved well-being among the EG compared to the CG at 3 months post intervention. One of the dimensions to assess well being includes:
  - anxiety and depression using the Hopkins Symptom Checklist-25 (values range from 1 to 4 per question with higher scores indicating worse outcomes)
General Wellbeing Measure | From enrollment until the end of 3 months post treatment follow up
  Improved well-being among the EG compared to the CG at 3 months post intervention. One of the dimensions to assess well being includes:
  - general wellbeing using the World Health Organization-5 questionnaire (values range from 0 to 5 per question with higher scores indicating better outcomes),
Self Efficacy Measure | From enrollment until the end of the intervention at 3 months post treatment
  Improved well-being among the EG compared to the CG at 3 months post intervention. One of the dimensions to assess well being includes:
  - self efficacy using the General Self-Efficacy Scale (values range from 1 to 4 per question, with higher scores indicating better outcomes)
Perceived Social Support Measure | From enrollment until the end of the intervention at 3 months post treatment
  Improved well-being among the EG compared to the CG at 3 months post intervention. One of the dimensions to assess well being includes:
  - perceived social support using the Multidimensional Scale of Perceived Social Support for Arab Women (values range from 1 to 7 per question with higher scores indicating better outcomes)

OTHER OUTCOMES:
Emotional Regulation Measure | From enrollement until 3 months post intervention delivery
  Improvement in key mediators in the EG compared to the CG at 3 months post intervention. Mediators will include emotional regulation measure through:
  - The Difficulties in Emotion Regulation Scale Short-Form (values range from 1 to 5, with higher scores indicating worse outcomes)
Interpersonal Communication Measure | From enrollment until 3 months post intervention
  Improvement in key mediators in the EG compared to the CG at 3 months post intervention. Mediators will include a communication measure through:
  - communication using the Interpersonal Communication Competency Scale (values range from 1 to 5, with higher scores indicating better outcomes)
Ways of Coping Measure | From enrollment until 3 months post intervention
  Improvement in key mediators in the EG compared to the CG at 3 months post intervention. Mediators will include emotional regulation measure through:
  - coping using the Revised Ways of Coping Checklist (values range from 0 to 3, with higher scores indicating better outcomes)

CONTACTS AND LOCATIONS:
Overall Officials: Shadi Saleh, PhD, Principal Investigator — Global Health Institute American University of Beirut; Lale Say, MD, Principal Investigator — World Health Organization
Locations (1):
- American University of Beirut, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No
Given the sensitive nature of the topic of this research, IPD will not be shared with other researchers. The studied population represents vulnerable individuals from refugee groups, and so ensuring confidentiality is necessary to keep in line with ethical guidelines and institutional policies, especially that IPD sharing was not communicated to AUB's IRB or to participants enrolled in the trial. Upon publication however, data can be made available as de-identified data to other researchers upon reasonable requests.

REFERENCES:
- [Derived] Sarieddine D, Chamseddine Z, Naal H, Dakdouki AE, Haidar GHA, Tamim H, Bosqui T, Fouad F, Ibrahim S, Sater ZA, Saleh S. Correlates of sexually transmitted infections among Syrian refugee women and girls in Lebanon: knowledge, symptoms, and health-seeking behaviors. BMC Womens Health. 2025 Oct 8;25(1):477. doi: 10.1186/s12905-025-04036-z. PMID 41063145
- See also: This link represents the SEEK trial study page on ELRHA's website. — https://www.elrha.org/project/self-efficacy-and-knowledge-to-improve-sexual-reproductive-health-and-wellbeing-in-humanitarian-settings-seek/